CLINICAL TRIAL: NCT03949881
Title: Cultured Autologous Oral Mucosa Epithelial Sheet for the Treatment of Bilateral Limbal Stem Cell Deficiency FEMJA for " Feuillet Epithélial de Muqueuse Jugale Autologue "
Brief Title: Cultured Autologous Oral Mucosa Epithelial Sheet for the Treatment of Bilateral Limbal Stem Cell Deficiency
Acronym: FEMJA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0032
Record Dates: First submitted 2019-05-13; First posted 2019-05-14 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Total Bilateral Limbal Cell Deficiency
Keywords: FEMJA transplantation; Epithelial jugal mucosa sheet; Limbal Stem-Cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FEMJA transplatation (Experimental): FEMJA epithelium is obtained by culturing oral mucosal epithelial cells without any need of support substrates, or carriers, and the transparent fabricated sheets show strong, rapid adhesion on corneal stroma in vivo, without any need for suturing.
  The cultivated oral mucosal epithelium will be directly grafted onto the corneal stroma. The sheet is grafted without suture onto the exposed stromal bed after removal of the conjunctiva and fibrosis from the cornea. The grafted corneal surface is then covered with a soft permanent contact lens for protection during healing (between 3 to 15 days, according to tolerance) If the stroma appears opaque because of deep stromal scars a corneal allograft will be performed 12 months after FEMJA transplantation.
  Interventions: Biological: FEMJA transplatation

INTERVENTIONS:
Biological: FEMJA transplatation — The cultivated oral mucosal epithelium will be directly grafted onto the corneal stroma. The sheet is grafted without suture onto the exposed stromal bed after removal of the conjunctiva and fibrosis from the cornea. The grafted corneal surface is then covered with a soft permanent contact lens for protection during healing (between 3 to 15 days, according to tolerance) If the stroma appears opaque because of deep stromal scars a corneal allograft will be performed 12 months after FEMJA transplantation.
  Other Names: Cultivated oral mucosal epithelium transplantation

SUMMARY:
Some severe ocular burns or other rare ocular pathologies can be associated with a total loss of corneal epithelial stem cells (i.e. Limbal Stem Cell Deficiency - LSCD), which leads to cornea invasion by the conjunctiva and a subsequent opacification. When LSCD is total and bilateral, both eyes are affected leading to full blindness and a poor quality of life, with a paradoxical photophobia that may be painful. Fewer than 100 patients bear this rare condition in France.

When patients suffer from total and bilateral LSCD, no treatment has been proven to provide clinical benefits: contralateral limbus is unavailable for autologous limbus graft or autologous limbal stem cells culture; allogeneic limbus graft requires immunosuppressive treatment leading to too important serious adverse effects compared to the expected benefit, and does not last long (< 2 years); and allogenic cornea transplantation is impossible since always rejected due to neovascularization.

A new way to treat these patients is to cultivate autologous corneal-like epithelium, and to graft it in order to restore transparency and to allow, if needed, a complementary corneal graft. Such an epithelium can be produced from autologous jugal mucosa cells. Epithelial jugal mucosa sheets transplantation has been assessed in a phase I/II clinical trial on 26 patients which showed that it is well-tolerated and effective but the culture technology used in this clinical trial is no longer available. A new enzymatic detachment process has been developed by the Hospices Civils de Lyon. Proof of concept was obtained from both in vitro and ex vivo studies: detachment with Collagenase at 0.5 mg/mL doesn't damage basement membrane proteins, so collagenase 0.5mg/mL-detached FEMJA were found to adhere, continue to ensure renewal of the differentiated epithelium 15 days after grafting onto an ex vivo porcine de-epitheliazed stroma model.

Considering these results, we aim to perform a clinical trial in order to evaluate tolerance and efficacy of the autologous jugal mucosa cell sheet (Feuillets Epithéliaux de Muqueuse Jugale Autologue - FEMJA) cultured with this innovative process.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* Signed and dated informed consent for participation in the study
* Total bilateral limbal stem-cell deficiency
* Caused by thermal or chemical burn, cornea transplantation, and other bilateral disorders of the ocular surface
* Severe loss of vision (<2/10 on decimal scale or/and EDTRS)
* The subject must be covered by a social security system

Exclusion Criteria

* Eye inflammation
* Strictly unilateral ocular affliction
* Acute systemic infection, objectified during consultation by the investigator and on the following paraclinical parameter: C Reactive Protein rate
* History of acute phase of ocular inflammation in the previous year
* History of neoplasic disease
* Glaucoma defined as intra ocular pressure (air tonometer and applanation tonometer) ≥ 22mmHg
* Total symblepharon (comprising eyelid aperture): impossibility to open the 2 eyes
* History of hyper sensibility or allergy to antibiotics or serum
* Women who are or may be pregnant or breastfeading
* Patients with any active infectious disease (HBV, HCV, HIV, HTLV-1 and syphilis)
* Patients who are otherwise ineligible for participation in the study in the opinion of the investigator.
* Delay of less than one year after chemical or thermal burns
* Person under judicial protection
* Contraindication related to anesthesia
* Contraindication to fluoresceine
* Oral mucosa tumor, pharynx or larynx tumor
* Fungal or viral infection of the ENT area
* Bacteria infection of the oral mucosa, pharynx or larynx.
* Hypersensitivity to ofloxacin (or other quinolone drugs), fluorometholone or betamethasone.
* Hypersensitivity to one of the excipients of the eye drops used: Monosodium phosphate, anhydrous disodium phosphate, polysorbate 80, sodium chloride, sodium edetate, polyvinyl alcohol, benzalkonium chloride, hydroxypropylmethylcellulose, hydrochloric acid, sodium hydroxide, lactose, cellulose, crospovidone, aspartam, magnesium stearate,
* Phenylketonuria
* Psychotic states not yet controlled by treatment;
* Vaccination with a live vaccine
* Bacterial, fungal, myco-bacterial infection of eye structures.
* Some evolving viral infections (including hepatitis, herpes, chickenpox, shingles) or other viral infections of the cornea or conjunctiva (except for a keratitis to Herpes zoster).
* Patients treated with Class IA or III antiarrhythmics, tricyclic antidepressants, macrolides and antipsychotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2031-05-13 (Estimated); Study Completion 2031-05-13 (Estimated)

PRIMARY OUTCOMES:
Number of patients with any improvement in visual acuity | 24 months after FEMJA transplantation
  Visual acuity measured at baseline (preoperative status) and 24 months after a jugal mucosa epithelial cell sheet transplantation (FEMJA transplantation), according to the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. ETDRS LogMAR tests allow measurement of very low visual acuity.

SECONDARY OUTCOMES:
Number of successful FEMJA transplantations | During 1 day of transplantation
  A success is defined by obtaining at least one FEMJA sheet that could be grafted without perforating it
Number of adverse events related to the procedure | Up to 24 months after FEMJA transplantation
  Adverse events related to the procedure; especially expected adverse events: inflammation, infection, and perforation.
Improvement in physical signs | 6 months, 12 months, 18 months and 24 months after FEMJA transplantation
  Any improvement from inclusion in physical signs measured with a slit lamp, in terms of: persistant epithelial defect; superficial punctate epithelial keratitis; and conjunctival epithelium on cornea.
Improvement in neovascularization | 6 months, 12 months, 18 months and 24 months after FEMJA transplantation
  Number of patients with a decrease in the number of vascular pediculus near the limbus and their activity, compared to inclusion.
Improvement in symptoms, i.e. functional signs | 6 months, 12 months, 18 months and 24 months after FEMJA transplantation
  Number of patients with an improvement in functional signs measured with Likert scales by self-reporting from the patient, in terms of: photophobia, eye dryness, and pain, compared to inclusion.
Corneal graft rejection | 24 months after FEMJA transplantation
  Among patients with secondary corneal graft, number of patients with graft rejection defined by intraocular pression (≥ 22mmHg) and significant increase in the thickness of the stroma of the cornea compared to the measured value just post graft on corneal topography.
Correlation between biological FEMJA characteristics and changes in visual acuity | 24 months after FEMJA transplantation
  FEMJA characteristics (extraction yield, percentage of proliferative epithelial cells) will be compared according to the clinical response for changes in visual acuity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology department, Edouard Herriot hospital, Hospices Civils de Lyon, Lyon, France